CLINICAL TRIAL: NCT05199129
Title: A Multi-center, Randomized, Double-blinded, Active-Controlled, Parallel, Phase III Study to Evaluate the Efficacy and Safety of HCP1904-3 in Essential Hypertension Patients
Brief Title: Clinical Efficacy and Safety Evaluation of HCP1904-3 in Essential Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-CHORUS-303
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Losartan; Chlorthalidone
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCP1904-3 (Experimental)
  Interventions: Drug: HCP1904-3; Drug: RLD2001-1
- RLD2001-1 (Active Comparator)
  Interventions: Drug: HCP1904-3; Drug: RLD2001-1

INTERVENTIONS:
Drug: HCP1904-3 — Take once daily for 8 weeks orally
Drug: RLD2001-1 — Take once daily for 8 weeks orally

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety of HCP1904-3 and RLD2001-1 alone in patients with essential hypertension inadequately controlled on RLD2001-1 monotherapy.

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-blinded, Active-Controlled, Parallel, Phase III Study to Evaluate the Efficacy and Safety of HCP1904-3 in Essential Hypertension patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 19 years of age
2. Patients who understands the process of clinical study and voluntarily signs a peer letter
3. Visit1: A person whose blood pressure measured in visit1 corresponds to the following conditions

   * Blood pressure medication taken patients: 130mmHg ≤ sitSBP<180mmHg, sitDBP<110mmHg
   * Blood pressure medication free patients: 140mmHg ≤ sitSBP<180mmHg, sitDBP<110mmHg
4. Visit2: 140mmHg ≤ sitSBP<180mmHg, sitDBP<110mmHg or if patients are in high risk group: 130mmHg ≤ sitSBP <180mmHg, sit DBP < 110mmHg

Exclusion Criteria:

1. Difference in mean value of blood pressure measured in both arms of more than 20mmHg in sitSBP or more than 10mmHg in sitDBP
2. Orthostatic hypotension with symptoms within 3months of visit 1
3. Secondary hypertensive patient or suspected to be
4. Uncontrolled diabetes mellitus(HbA1c > 9%) or type I diabetes mellitus
5. Active gout or hyperuricemia (uric acid ≥ 9mg/dL)
6. Severe heart disease or severe neurovascular disease
7. Severe or malignant retinopathy
8. Clinically significant hematological finding
9. Severe renal diseases (eGFR<30mL/min/1.73m2)
10. Severe hepatopathy or active hepatopathy (AST or ALT normal range ≥ 3 times)
11. Hypokalemia or Hyperkalemia(K<3.5mmol/L or K ≥ 5.5mmol/L)
12. Hyponatremia or Hypernatremia(Na<135mmol/L or Na ≥ 155mmol/L)
13. Hypercalcemia
14. History of malignancy tumor
15. History of autoimmune disease
16. History of alcohol or drug abuse
17. Positive to pregnancy test, nursing mother, intention on pregnancy
18. Considered by investigator as not appropriate to participate in the clinical study with othe reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure(mmHg) | Week 8

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure(mmHg) | Week 4
Change from baseline in mean sitting diastolic blood pressure(mmHg) | Week 4,8
Change from baseline in mean pulse blood pressure(mmHg) | Week 4,8
Target blood pressure reach rate(%) | Week 4,8
Blood pressure responder rate(%) | Week 4,8

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea